CLINICAL TRIAL: NCT04052802
Title: The Efficacy Of A Bioactive Resin Material Used As A Fissure Sealant As Compared To A Conventional Resin Regarding Its Retention, Marginal Integrity And Prevention Of Lesion Progression. A Randomized Clinical Study
Brief Title: Compariing a Bioactive Resin Material Used As A Fissure Sealant To A Conventional Resin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Khaled Mostafa, Researcher, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 812014
Record Dates: First submitted 2019-08-05; First posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Demineralization, Tooth; Demineralization, Fissure; Non-Cavitated Caries
MeSH Terms: conditions — Tooth Demineralization

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bioactive resin (Giomer) (Experimental): This group of patients will receive a bioactive resin "Beautifil flow plus X (Shofu Dental)" for treatment of their demineralized fissures
  Interventions: Other: Fissure sealing
- Conventional resin (Experimental): This group of patients will receive a conventional resin "Filtek Z350xt Flowable composite (3M ESPE)" for treatment of their demineralized fissures
  Interventions: Other: Fissure sealing

INTERVENTIONS:
Other: Fissure sealing — The materials will be applied to the demineralized fissures as stated in manufacturer's instructions

SUMMARY:
The aim of this study is to investigate the retention, marginal integrity and potential to prevent lesion progression of a bioactive resin material compared to a conventional resin-based flowable composite during management of initial carious lesion in adult population over an 18 months period.

DETAILED DESCRIPTION:
Bio-active resin materials aim to possess the mechanical properties of resin materials in terms of higher wear resistance and dimensional stability over time. They also aim to mimic the biological activity of glass ionomers in terms of ion recharge and release. These new bio-active resin materials, with their lower particle size and better adaptability and polishability, might offer a substantial addition as fissure sealants if they fulfil the requisities satisfactory mechanical properties of resins and of ion recharge and release of glass ionomers.

The study will be conducted on demineralized fissures of permanent molars by application of a newly introduced giomer in one group while the other group will recieve a conventional resin material where they will be assessed for retention, marginal integrity and caries progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with good oral hygiene
* Co-operative patients with initially demineralized fissures in permanent molars of the maxilla or mandible

Exclusion Criteria:

* Medical Problems or Pregnancy
* Lack of patient's approval and compliance
* Presence of abnormal oral, medical, or mental condition
* Known allergy of resin-based materials
* Previous placements of sealants or restorations
* Bruxism or mal-occlusion

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-08-30 (Estimated); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Retention | 18 months
  The sealing materials will be assessed for complete, partial or no retention. The assessment will be carried out by visual and tactile assessments and calculated as a percentage of the total sample.

SECONDARY OUTCOMES:
Marginal integrity | 18 months
  The materials margins will be assessed for their marginal seal using FDI criteria using a WHO probe. Scoring will be made from 1-5 by FDI criteria then statistically analyzed
Caries progression | 18 months
  The demineralized fissures will be monitored for caries arrest or progression. The assessment will be made by ICDAS II criteria comparing the scores from baseline.

IPD SHARING:
Plan to Share IPD: No
The data will be assessed collectively for ll participants and statistically analyzed and published with the results. Other data can be provided apon request if ethically approved.